CLINICAL TRIAL: NCT04874987
Title: Impact of Simulation Based Learning on Gender, and Equity Dynamics Among Interhealth Professionals at Selected Institutions in Sub Saharan Africa
Brief Title: Impact of Simulation Based Learning on Gender, and Equity Dynamics Among Inter-health Professional Teams
Acronym: Sim-Gender
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mbarara University of Science and Technology (Other)
Collaborators: University of Calgary (Other); The ELMA Foundation (Other); Alberta Children's Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/MUST-3/SIM-II
Record Dates: First submitted 2021-04-18; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Simulation-based Methodology
Keywords: Simulation based learning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Simulation based learning with Advocacy inquiry and ladder of influence — Simulation scenarios based on identified gender and equity gaps. We will explore experiences of male and female participants, and inter-professional simulation participants (e.g nurses and doctors, medical and nursing students) post intervention exposure on their role and experiences in simulated sessions and clinical care experiences
  Other Names: Gender sensitive simulation based learning

SUMMARY:
At Mbarara University of Science and Technology and partner sites, the investigators will explore the role of simulation in gender and equity. African societies are largely patriarchal, and this spills over into professional practice and medical education. Simulation methodology is at risk of suffering from a patriarchal dominance. The male dominance has potential to introduce power relationships between men and women learners in a scenario setting and between physicians and nurses. In the presence of such power differentials, the less dominant party could develop a "culture of silence," fail to take decisions on issues that affect them or their patients, fail to talk about these issues and take appropriate action.

DETAILED DESCRIPTION:
To address the challenges of gender and equity: 1) the investigators will teach Advocacy Inquiry (AI) and the ladder of inference (LoI) as conversational strategies for all simulation faculty members to explore participant frames of action and thought processes, 2) the investigators will design and expose participants to simulated scenarios with embedded gender and or inter-professional power differentials, 3) study the effect of AI, the LoI and debriefed gender and equity scenarios on participant engagement strategies during gender and inter-professional conflict situations.

The Ladder of Influence allows facilitators select some data / observation, add interpretation, draw conclusions and take action. Though the Ladder of influence is a powerful approach to exploring situations, its prone to challenges if users jump to conclusions quickly without being curious about what alternative interpretations of the observed data / action could be. AI uses the "show", "think" and "wonder" as a strategy to slow facilitators from jumping up the LoI to draw conclusions before exploring learner perspectives. AI and the LoI in combination encourage self-reflection and good judgment. The investigators will deliberately encourage simulation teams to have both males and females and inter-professional with opportunities for team leaders to vary with both sex and profession.

ELIGIBILITY:
Inclusion Criteria:

* Medical students
* Faculty members in the Faculty of Medicine
* Based at Mbarara University, Lira University, Busitema University, or Muni University

Exclusion Criteria:

* Medical students and faculty outside the participating Universities
* Non-medical students
* Faculty not based in the Faculties of Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical students, faculty members involved in delivery of scenario execution
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Gender and inter-professional conflicts in simulation | Change in conflicts 24 months after introduction of simulation based techniques
  Frequency of gender and inter-professional conflicts reported in simulation session and or clinical care spaces during debriefing sessions

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No
Data will not be shared given the private nature (involves videos)